CLINICAL TRIAL: NCT00697606
Title: Randomized Double-Blind Controlled Study to Determine if Seprafilm® Reduces Adhesions After Primary Cesarean Section
Brief Title: Seprafilm® for Prevention of Adhesions at Repeat Cesarean
Acronym: SPARC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Abington Memorial Hospital (Other)
Responsible Party: Principal Investigator, David Peleg, MD, Principle Investigator, Abington Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Study #08-032
Record Dates: First submitted 2008-06-12; First posted 2008-06-16 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Adhesion Formation After Primary Cesarean Delivery
Keywords: Seprafilm®; cesarean; adhesions; primary; repeat
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Seprafilm®
  Interventions: Device: Seprafilm®
- B (Sham Comparator): Control
  Interventions: Other: Control

INTERVENTIONS:
Device: Seprafilm® — Seprafilm® placed at time of primary cesarean
  Arms: A
Other: Control — no Seprafilm® used at primary cesarean
  Arms: B

SUMMARY:
Adhesion formation is a result of abdominal and pelvic surgery and is a cause of such diseases as chronic pain syndrome, bowel obstruction and infertility. Both patients and surgeons suffer when adhesions are encountered, since the surgery becomes more intense, lengthy, and complicated. Seprafilm® has been shown to limit the formation of adhesions in gynecologic and abdominal surgery. Limited data is available on the effectiveness of Seprafilm® in the prevention of abdominal wall and pelvic adhesions at the time of cesarean section. Adhesions at the time of repeat cesarean make the surgery frustrating and complex, with difficult lysis of adhesions being the cause of morbidities such as bladder damage, increased blood loss, and longer operating times. The objective of this definitive project is to define the extent of reduction of adhesion formation of Seprafilm® when used at the time of primary cesarean section. Women undergoing primary cesarean section will be randomized for Seprafilm® application, and the incidence and grade of adhesions at repeat cesarean will be determined.

DETAILED DESCRIPTION:
This is a prospective randomized double-blinded study. Patients will be randomized prior to primary cesarean section to either the study arm (Seprafilm® placement) or control arm (nothing placed). Seprafilm® will be placed over the repaired uterine incision and over the anterior aspect of the uterus prior to closure of the fascia (2 to 3 sheets per patient). Randomization will be by opaque envelops containing group assignment.

Participants and surgeons will be blinded to group designation at the time of repeat cesarean. The surgeon will be asked to grade the adhesions at the time of repeat cesarean.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women after 24 weeks' gestation.
2. First cesarean delivery.
3. Age > 18 years.
4. Cesarean to be performed by a participating surgeon.
5. Non-closure of the visceral or parietal peritoneum.

Exclusion Criteria:

1. Any prior abdominal surgery including prior cesarean, laparoscopy, appendectomy, cholecystectomy or any uterine adnexal or bowel surgery.
2. Clinical diagnosis of chorioamnionitis.
3. Women having tubal ligation at the time of primary cesarean.
4. Inability to obtain informed consent.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 450 (Actual)
Dates: Start 2008-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To determine if Seprafilm® decreases the incidence of adhesion formation by 50% after primary cesarean. | at repeat cesarean

SECONDARY OUTCOMES:
To determine to what extent Seprafilm® decreases the incidence of adhesion formation. | at repeat cesarean
To determine the incidence of adhesion formation during repeat cesarean delivery. | at repeat cesarean
To evaluate complication rates in those with Seprafilm® versus those without during repeat surgery by examining length of operating times, blood loss, bladder injuries, and Apgar scores | at repeat cesarean
To determine the incidence of fertility issues in women having Seprafilm® placed during primary cesarean delivery versus those not having Seprafilm® placed. Participating women will be contacted by telephone every 4 months. | ongoing during trial

CONTACTS AND LOCATIONS:
Overall Officials: Amy Mackey, MD, Principal Investigator — Abington Memorial Hospital; Mark Shahin, MD, Principal Investigator — Abington Memorial Hospital; Richard Latta, MD, Principal Investigator — Abington Memorial Hospital; David Peleg, MD, Principal Investigator — Abington Memorial Hospital
Locations (1):
- Abington Memorial Hospital, Abington, Pennsylvania, United States